CLINICAL TRIAL: NCT01801722
Title: Using NT-proBNP to Detect Chronic Heart Failure in Patients With Chronic Obstructive Pulmonary Disease.
Acronym: NT-proBNP
Status: Completed | Type: Observational
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Elzbieta Kaszuba, PhD student, Lund University
Other Study IDs: 502008; DN50/2008 (Other: Ethics committee at Lund university)
Record Dates: First submitted 2013-02-25; First posted 2013-03-01 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NT-proBNP,ejection fraction ,COPD stage.: The group comprised 25 women (47%) and 28 men (53%). The mean age was 75.4 years (SD 7.9), 76.3 (SD 7.6) for men and 74.4 (SD 8.2) for women.

SUMMARY:
The aim of the present study was to evaluate if the analysis of NT-proBNP might be used as an initial step for the diagnosis of chronic heart failure in patients with COPD in primary health care, and to select patients for a further examination by echocardiography.

DETAILED DESCRIPTION:
Patients with a confirmed diagnosis of COPD were examined regarding chronic heart failure.

1. An interview regarding symptoms: breathlessness, orthopnoea, night cough, nocturia, walking distance.
2. Physical examination: weight and height, heart and lung auscultation, blood pressure measurement after 5 minutes' rest in the sitting position and the presence of peripheral oedema.
3. Electrocardiography.
4. Natriuretic peptide- NT-proBNP (Immulite 2500, Siemens Healthcare Diagnostics AB Sweden).
5. Patients with the NT-proBNP level of > 1200 pg/ml were referred for echocardiography to assess left ventricular function.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older with the following diagnosis codes according to International Statistical Classification of Diseases and Related Health Problems - Tenth Revision:J44 (COPD) and J41, J42 (chronic bronchitis) registered during the period 1 January 2008-16 April 2008 according to the electronic patient record.

Exclusion Criteria:

* Impaired cognitive function and/or anticipated difficulties in carrying out spirometry due to immobility,
* psychiatric disorders or terminal illness.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older with a registered diagnosis of COPD.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with elevated NT-proBNP. | 3 months
  NT-proBNP has taken only once in each patient without follow up follow up. Three months was a period when we collected data from all participants.

SECONDARY OUTCOMES:
Percentage of patients with abnormal left ventricular function assessed by echocardiography. Association between elevated NT-proBNP and symptoms, signs and electrocardiography. | 3 months
  Echocardiography was performed once in each referred patient. Three months was a period of data collection.

CONTACTS AND LOCATIONS:
Overall Officials: Elzbieta Kaszuba, PhD student, Principal Investigator — Lund University
Locations (1):
- Primary health care center., Olofström, Blekinge County, Sweden